CLINICAL TRIAL: NCT06641882
Title: Retrospective Chart Review of Patients With Acanthamoeba Keratitis Who Have Received 0.8 mg/ml Polihexanide as Part of a Compassionate Use Program: A Non-interventional Study With Secondary Use of Data
Brief Title: Retrospective Chart Review of Patients With Acanthamoeba Keratitis Who Have Received 0.8 mg/ml Polihexanide
Status: Completed | Type: Observational
Sponsor: SIFI SpA (Industry)
Responsible Party: Sponsor
Other Study IDs: 057/SI
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-07

CONDITIONS: Acanthamoeba Keratitis
MeSH Terms: conditions — Acanthamoeba Keratitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This will be a non-interventional study with secondary use of data. The study will be a site-based retrospective review of medical chart of patients with AK who initiated and completed a treatment with 0.8 mg/ml polihexanide as part of a compassionate use program. Patientlevel data will be abstracted from medical chart of eligible patients at participating sites and imputed in an electronic case report form (eCRF). Baseline (Time 0) is the date of initiation of 0.8 mg/ml polihexanide. The study period is the period from T0 to the end of treatment. The clinical outcome needs to be confirmed at least 30 days after the conclusion of the treatment.

DETAILED DESCRIPTION:
Acanthamoeba keratitis (AK) is an ultra-rare potentially devastating ocular infection that occurs primarily in contact lens wearers. The estimated incidence in Europe varies between 1 and 3 cases/million people per year. AK is caused by a ubiquitous free-living protozoan that is present in air, soil, dust, fresh water, seawater, and bottled water. The amoebic organism exists both as dormant cysts and active trophozoites. The cysts are highly resilient and can withstand a wide variety of physical conditions and drugs which makes medical treatment of AK both difficult and protracted. If left untreated, the cure rate is low with most patients needing keratoplasty and some of them requiring enucleation. There is currently no approved pharmacological treatment for AK. Available treatment options are represented by off-label antiseptic products which are either imported or compounded, the most used being biguanides (polihexanide-PHMB- or chlorhexidine), given alone or in combination with a diamidine (propamidine or hexamidine). The actual reported medical cure rate with no surgery is approximately 60%; in addition almost 50% of patients have a poor outcome, defined as a poor visual acuity and/or necessity of ocular surgery. Polihexanide 0.8 mg/ml, an eye drops solution developed and manufactured by SIFI SpA (Italy), has the potential to become the first treatment approved for the treatment of AK. Its efficacy and safety were demonstrated in the pivotal clinical study 043/SI (EUDRACT no. 2016-001823-30; ClinicalTrials.gov: NCT03274895), in which the mean (95% IC) cure rate with no surgery was 84.8% (73.9-92.5) with a median (95% IC) time-to-cure of 146 (94-217) days. In addition, no major safety issues were observed during the trial. A positive opinion from the Committee for Medicinal Products for Human Use at EMA is expected in Q2/2024. Polihexanide 0.8 mg/ml has been made available in Italy by SIFI S.p.A. through a compassionate use program (CUP) since November 2022 (Compassionate use program, version 1.1-ITA-Aug 11, 2022). As of December 2023, the treatment with 0.8 mg/ml polihexanide was approved for 71 patients with AK. SIFI prepared this protocol to conduct a retrospective medical chart review of patients which already completed the treatment with 0.8 mg/ml polihexanide as part of the CUP. The expected number of evaluable patients is 40. According to the European Network of Centres for Pharmacoepidemiology and Pharmacovigilance (ENCePP) this will be a Non-Interventional Study (as defined in the Directive 2001/20/EC) with secondary use of data. The protocol was prepared following the good practices report of the ISPE/ISPOR task force.

The expected contribution from this study will be to expand patient's exposure to polihexanide 0.8 mg/ml and provide further information on its effectiveness and safety when used in the clinical practice compared with the findings observed in the pivotal clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Age >14 years.
* Clinical signs and symptoms consistent with AK.
* Identification of Acanthamoeba (diagnostic confirmation of AK) by at least one of the allowed techniques as:

  * Confocal Microscopy
  * PCR,
  * Identification by microbiological culture or cytological smear.
* Accept to sign the informed consent.

Additional inclusion criteria:

* Inclusion in the compassionate use program from 1st December 2022 to 31st December 2023 (date of approval by the local Ethics Committee).
* Treatment with 0.8 mg/ml polihexanide.
* End of treatment with 0.8 mg/ml polihexanide.
* Medical chart available at clinical site.

Exclusion Criteria: None

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects included in the study will be patients who have received 0.8 mg/ml polihexanide through the CUP. Clinical sites with at least 3 patients in the CUP will be selected.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-09-30 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
To describe the effectiveness of 0.8 mg/ml polihexanide as measured by the proportion of patients cured over time, between baseline (T0) and end of study period. | The study period is the period from T0 to the end of treatment (Up to 52 weeks)
  The outcome of interest will be the medical cure defined as the presence of an intact corneal epithelium, no or mild signs of ocular inflammation and no surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Karl Knutsson, MD, Principal Investigator — San Raffaele Scientific Institute
Locations (10):
- Italy (10):
  - ASST Spedali Civili, Brescia, Brescia
  - SOD Oculistica Azienda Ospedaliero Universitaria Careggi, Florence, Italy
  - IRCCS Ospedale San Raffaele, Milan, Italy
  - AZIENDA ULSS 3 Serenissima-UOC Oculistica, Venice, Italy
  - Policlinico G.Martino, Messina, Messina
  - ASST Fatebenefratelli Sacco, Milan, Milano
  - Policlinico S. Matteo, Pavia, Pavia
  - Policlinico TorVergata, Rome, Rome
  - Policlinico Universitario Campus Biomedico, Rome, Rome
  - Azienda Ospedaliera Universitaria Verona, Verona, Verona